CLINICAL TRIAL: NCT03359564
Title: Microendoscopic Lumbar Discectomy: A Prospective Study of 100 Cases
Brief Title: Microendoscopic Lumbar Discectomy: A Study of 100 Cases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, guochen, department of spinal surgery, Peking University People's Hospital
Other Study IDs: MED007
Record Dates: First submitted 2017-11-26; First posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Lumbar Disc Herniation
Keywords: Lumbar Disc Herniation; Micro Endoscopic Discectomy
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- micro endoscopic discectomy: the patients with lumbar disc herniation
  Interventions: Procedure: micro endoscopic discectomy

INTERVENTIONS:
Procedure: micro endoscopic discectomy — the patients receive micro endoscopic discectomy surgery therapy

SUMMARY:
Evaluate the outcome of micro endoscopic discectomy (MED) by tubular retractors on safety and efficacy of the technique.

DETAILED DESCRIPTION:
Evaluate the outcome of micro endoscopic discectomy (MED) by tubular retractors on safety and efficacy of the technique.Patients who underwent surgery for herniated disc using the tubular retractors. The results were evaluated by using VAS (Visual Analog Scale 0-5) for back and leg pain and ODI (Oswestry Disability Index). Patients were followed up at intervals of 1 week, 6 weeks, 3 months, 6 months, 12 months and 2 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least 6 weeks of conservative treatment with positive nerve root tension signs, radicular pain
* Patients are diagnosed with lumbar disc herniation by MRI
* Patients who underwent surgery for herniated disc using the tubular retractor

Exclusion Criteria:

* Patients with large central disc herniation, chronic discogenic pain, discitis, multi-level disease, presence of instability or history of lumbar surgery

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent surgery for herniated disc using the tubular retractor
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index | 2 years after operation
  The efficacy of surgery were evaluated by using Oswestry Disability Index.

SECONDARY OUTCOMES:
Oswestry Disability Index | preoperative evaluation and 1 week, 6 weeks, 3 months, 6 months, 12 months after operation
  The efficacy of surgery were evaluated by using Oswestry Disability Index.
Visual Analog Scale | preoperative evaluation and 1 week, 6 weeks, 3 months, 6 months, 12 months and 2 years postoperative follow-up
  The efficacy of surgery were evaluated by using Visual Analog Scale for back and leg pain.

CONTACTS AND LOCATIONS:
Overall Officials: GUO chen, bachelor, Principal Investigator — department of spinal surgery,PekingUPH

IPD SHARING:
Plan to Share IPD: Undecided